CLINICAL TRIAL: NCT03384472
Title: Integrating Genetic Epidemiology as an Intensified Surveillance Tool Into the National Centre for Parasitology, Entomology and Malaria Control of Cambodia
Brief Title: Malaria Genetic Surveillance in Cambodia
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); National Centre for Parasitology, Entomology and Malaria Control, Cambodia (Other)
Responsible Party: Sponsor
Other Study IDs: BIOINF1601
Record Dates: First submitted 2016-08-22; First posted 2017-12-27 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2017-12

CONDITIONS: Parasitology; Entomology; Malaria
Keywords: Malaria Genetic Surveillance; Cambodia
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dried blood spots (DBS) will be obtained through finger prick blood sampling from patients, with three blood spots on one piece of filter paper being obtained from each patient. Each blood spot will contain ~20µl of blood, for a total of ~60µl of blood being collected from each patient for the study.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to determine the prevalence and geographical distribution of antimalarial drug resistance-linked genetic mutations in clinical P. falciparum infections in Cambodia

DETAILED DESCRIPTION:
This is a prospective observational study of patients with clinical Plasmodium falciparum infection using parasite DNA from point-of-care fingerprick dried blood spot samples as well as a short survey on patient demographics, employment, travel, and mobile phone use to study P. falciparum parasite genotypes, population characteristics, and gene flow patterns.

On inclusion in the study and before standard treatment is administered, dried blood spots (DBS) will be obtained through fingerprick blood sampling from patients, with three blood spots on one piece of filter paper being obtained from each patient. Each blood spot will contain ~20µl of blood, for a total of ~60µl of blood being collected from each patient for the study.

In order to have a greater understanding of the possible sites of malaria transmission and to relate genetic diversity to geographic location, patients or their parents/guardians will also be asked a short set of questions on demographics, their places of residence and work, recent mobile phone use, and their history of travel in the last 2 months. As some of this information can be sensitive, during the consent process the patient will be given the option of not providing some or all of this information without needing to provide a reason. This is explained on the patient information sheet. For those who do not want to provide information, this will be documented in the survey form. A duplicate of the sample barcode will be placed on this same form, so the information therein can be matched with the relevant blood spot and its related genetic data, while retaining sample anonymity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >6 months of age
* P. falciparum malaria as confirmed by positive rapid diagnostic test or asexual forms of P. falciparum on blood smear microscopy (may be mixed with non-falciparum Plasmodium species)
* Written informed consent by patient, parent/guardian, or legally authorised representative to participate in the study

Exclusion Criteria:

• None

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients > 6 months of age with P. falciparum malaria who present to village malaria workers and health centres in Stung Treng and Ratanakiri provinces in Cambodia are the target study population. 2014 data suggest this could amount to up to 7,000 patients per year. All study participants must satisfy the applicable inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Annual maps and reports on the prevalence of drug resistance-linked genetic mutations in P. falciparum parasites in Cambodia | up to 12 months

SECONDARY OUTCOMES:
Population structure of P.falciparum parasites | up to 12 months
  By using population genetics and clustering techniques, such as Principal Component Analysis and phylogeny
Gene flow patterns of P. falciparum malaria parasites in Cambodia | up to 12 months
Likely geographic origin of P. falciparum malaria parasites in Cambodia | up to 12 months

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data recorded in the CRFs will be shared via open access online repositories as per the requirements of the journal in which the results of the study are published.

REFERENCES:
- [Result] Jacob CG, Thuy-Nhien N, Mayxay M, Maude RJ, Quang HH, Hongvanthong B, Vanisaveth V, Ngo Duc T, Rekol H, van der Pluijm R, von Seidlein L, Fairhurst R, Nosten F, Hossain MA, Park N, Goodwin S, Ringwald P, Chindavongsa K, Newton P, Ashley E, Phalivong S, Maude R, Leang R, Huch C, Dong LT, Nguyen KT, Nhat TM, Hien TT, Nguyen H, Zdrojewski N, Canavati S, Sayeed AA, Uddin D, Buckee C, Fanello CI, Onyamboko M, Peto T, Tripura R, Amaratunga C, Myint Thu A, Delmas G, Landier J, Parker DM, Chau NH, Lek D, Suon S, Callery J, Jittamala P, Hanboonkunupakarn B, Pukrittayakamee S, Phyo AP, Smithuis F, Lin K, Thant M, Hlaing TM, Satpathi P, Satpathi S, Behera PK, Tripura A, Baidya S, Valecha N, Anvikar AR, Ul Islam A, Faiz A, Kunasol C, Drury E, Kekre M, Ali M, Love K, Rajatileka S, Jeffreys AE, Rowlands K, Hubbart CS, Dhorda M, Vongpromek R, Kotanan N, Wongnak P, Almagro Garcia J, Pearson RD, Ariani CV, Chookajorn T, Malangone C, Nguyen T, Stalker J, Jeffery B, Keatley J, Johnson KJ, Muddyman D, Chan XHS, Sillitoe J, Amato R, Simpson V, Goncalves S, Rockett K, Day NP, Dondorp AM, Kwiatkowski DP, Miotto O. Genetic surveillance in the Greater Mekong subregion and South Asia to support malaria control and elimination. Elife. 2021 Aug 10;10:e62997. doi: 10.7554/eLife.62997. PMID 34372970
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34372970/